CLINICAL TRIAL: NCT01112176
Title: Effect of Heart Rate on Left Ventricular Performance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: David S. Blondheim, MD, Hillel Yaffe Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 013-10-HYMC-CTIL
Record Dates: First submitted 2010-04-13; First posted 2010-04-28 (Estimated); Last update posted 2010-04-28 (Estimated); Status verified 2010-04

CONDITIONS: Myocardial Function; Myocardial Strain
Keywords: Strain; Ejection fraction; Diastolic function
MeSH Terms: conditions — Sprains and Strains

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Increase in paced heart rate — The pacing rate will be increased by 10 bps at every stage

SUMMARY:
The current study is aimed at determining the normal response to increasing heart rates. For this purpose, atrial pacing will be used to increase heart rate.

DETAILED DESCRIPTION:
Participants will be patients with pacemakers and normal A-V node conduction with a possibility for right atrial pacing mode.

Detailed Echo studies will be performed at baseline. Echo studies will be repeated at each pacing stage, stages defined as 10 bpm increments in paced heart rate. Each stage will last 2-3 min or as long as it takes to record the echo study. Heart rate will be increased to 85% of predicted heart rate for age or at to appearance of signs of ischemia.

Hemodynamic parameters will be recorded and segmental longitudinal strain will be calculated (as well as other Echo data), for each stage.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with AAI or DDD pacemaker with intact AV nodal conduction that can be set to work in AAI mode.
2. Stable rhythm (either sinus or paced).
3. Good quality baseline echo.
4. Able and willing to sign Informed Consent Form.

Exclusion Criteria:

1. Prior heart failure or ischemic heart disease.
2. Severe valvular lesions.
3. Severe pulmonary hypertension.
4. Known intolerance to rapid pacing.
5. Multiple extrasystoles (more than 1 per echo or monitor screen).
6. Age over 70.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-04; Primary Completion 2012-04 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
Segmental Strain | approx. 20 minutes
  Segmental Strain by speckle tracking method will be calculated for every stage of each study.

SECONDARY OUTCOMES:
LV function | Approx. 20 minutes
  Parameters of systolic and diastolic function will be calculated at each stage.

CONTACTS AND LOCATIONS:
Overall Officials: David S. Blondheim, MD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hille Yaffe Medical Ceter, Hadera, Israel, Israel